CLINICAL TRIAL: NCT00552916
Title: Functional Electrical Stimulation (FES)-Assisted Walking: Enhancement of Voluntary Walking Function Among Persons With Severe Hemiplegia Post-Stroke
Brief Title: Functional Electrical Stimulation (FES) Assisted Walking: Enhancement of Walking Function After Stroke
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Dr. Milos R. Popovic, Toronto Rehab: Lyndhurst Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SRA 5973; NCT00538837 (obsolete NCT alias)
Record Dates: First submitted 2007-11-01; First posted 2007-11-02 (Estimated); Last update posted 2008-08-20 (Estimated); Status verified 2008-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Participants will be randomized to either an intervention arm where they will receive 'true' FES and the other control arm where they will receive 'false' FES. The sham group will receive 'false' FES.
  Interventions: Device: Compex Motion Stimulator
- 2 (Other): The intervention group will receive 'true' FES
  Interventions: Device: Compex Motion Stimulator

INTERVENTIONS:
Device: Compex Motion Stimulator — 'True' Functional Electrical Stimulation Assisted Walking
  Arms: 2
Device: Compex Motion Stimulator — 'False' FES
  Arms: 1

SUMMARY:
The purpose of this study is to determine if a form of exercise,known as electrical stimulation can improve walking function and other important health outcomes. The hypothesis is that electrical stimulation can enhance the ability to walk for stroke survivors who are unable to walk on their on their own.

DETAILED DESCRIPTION:
A stroke is a devastating life event, that can result in permanent disability. Many people who survive a stroke will experience paralysis on one side of their body. The muscles in one leg may become weaker or stiff to the point that the person can barely walk. Functional electrical stimulation (FES) is an intervention that applies short current pulses to muscles and causes them to contract. Previous work done by our team has used FES in the spinal cord injured population to help restore functions such as walking and grasping by contracting groups of paralyzed muscles in an orchestrated manner. This study seeks to explore whether a thrice weekly FES-assisted walking intervention for a 8 week period can stimulate or improve walking ability in individuals with severe lower extremity paralysis secondary to a stroke. This will subsequently promote opportunities for enhanced social participation and quality of life i.e. enhanced balance, increased independence of activities of daily living etc. for stroke consumers. Comparison: 40 individuals with severe hemiplegia will be randomized to either a thrice weekly control (false) FES training regimen OR a thrice weekly intervention (true) FES training regimen. Prior to randomization, participants will be stratified according to their ability to ambulate (walk). This study will determine if FES can improve or enhance walking ability associated with stroke after 8 weeks of training, and after 4-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegic stroke at least 12 months prior to joining the study.
* Age 65 years or greater.
* Ability to follow instructions and to devote his/her attention to therapy.
* Ability to understand instructions in English and able to provide informed consent.

Exclusion Criteria:

* Severe difficulties with attention such that informed consent cannot be obtained, or that safety or communication would be comprised.
* Ability to walk more that 10 meters during a two minute walk with an average speed greater than 0.8 m/s.
* The presence of skin rashes, allergies or bruises where electrodes would be placed.
* History of seizures, edema in paralyzed limbs or co-morbidities such as Parkinson's Disease, cancer or osteoarthritis to be confirmed by attending physiatrist.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-10; Primary Completion 2010-10 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
The ability of FES-Assisted Walking to stimulate or improve walking ability using a dichotomous outcome i.e. yes/no stimulation or improvement of walking ability on a two-minute walk test. | Test performed weekly during 8-week period as well as at 2 month and 6 month time point.

SECONDARY OUTCOMES:
Assessment of balance by completing four tests i.e. move from a seated to a standing position, completion of activities of daily living tasks such as moving from a bed to a wheelchair, standing with eyes opened and closed. | Baseline, 2 month and 6 month period.
Bone density at hip, spine, proximal tibia and distal femur using dual-energy xray absorptiometry | Baseline, 2-month and 6-month
Assess functional abilities by performing various tasks using our leg and foot as well as your ability to perform functional tasks such as eating, grooming and bathing. | Baseline, 2-month and 6-month time points.

CONTACTS AND LOCATIONS:
Overall Officials: Milos R Popovic, PhD, Principal Investigator — University of Toronto
Locations (1):
- Toronto Rehabilitation Institute: Lyndhurst Centre, Toronto, Ontario, Canada